CLINICAL TRIAL: NCT01759628
Title: The Effect of Helicobacter Pylori Eradication on Liver Function Tests in Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: Helicobacter Pylori Eradication in Subjects With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Kashan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Raika Jamali, MD, Assistant Professor of Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91138 - KAUMS
Record Dates: First submitted 2012-12-20; First posted 2013-01-03 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Steatohepatitis,; Helicobacter pylori,; Insulin resistance,; Alanine aminotransferase,; Aspartate aminotransferase,
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle modification (No Intervention): Obtaining ideal body weight by calorie restriction diet and programmed physical activity
- H.pylori eradication (Experimental): H.pylori eradication by quadruple antibiotic therapy for two weeks plus obtaining ideal body weight by calorie restriction diet and programmed physical activity
  Interventions: Drug: H.pylori eradication

INTERVENTIONS:
Drug: H.pylori eradication — The regimen consists of Omeprazole (20 mg/BD)+ Amoxicillin (1 g/day)+ Bismuth subcitrate (240 mg/BD)+ Azithromycin (500 mg/BD)for two weeks
  Other Names: Helicobacter pylori treatment
  Arms: H.pylori eradication

SUMMARY:
The aim of study was to evaluate the effect of helicobacter pylori eradication on liver function tests, lipid profile, homeostasis model assessment-IR (HOMA-IR) index, and anthropometric measurements (body mass index and waist circumference)in subjects with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Helicobacter pylori (HP) antigens have been found in the liver of individuals with benign and malignant liver diseases. The role of HP in the pathogenesis of non-alcoholic fatty liver disease (NAFLD) is controversial.

This randomized double blind clinical trial was performed in dyspeptic patients with positive antibody to HP and the evidence of fatty liver in ultrasonography. After excluding other causes, participants with persistent elevated serum aminotransferase levels were presumed to have NAFLD. Those with NAFLD liver fat score greater than (-0.64) and positive urea breath test (UBT) were enrolled. They were randomly assigned to lifestyle modification alone or lifestyle modification plus HP eradication groups. Quadruple therapy (omeprazole, amoxicillin, bismuth subcitrate, and clarithromycin) for HP eradication was performed in two weeks. HP eradication was documented by UBT. Fasting serum glucose, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, triglyceride, cholesterol, high and low-density lipoprotein, HOMA-IR, and anthropometric measurements (body mass index and waist circumference) were checked at baseline, eight weeks, and twelve weeks from the beginning of study.

ELIGIBILITY:
Inclusion Criteria:

* Dyspeptic patients with positive antibody to H.pylori and persistent elevated aminotransferase levels with the evidence of fatty liver in ultrasonography, who were referred to a gastroenterology clinic

Exclusion Criteria:

* Alcohol use (more than 20 gram per day in men and 10 gram per day in women per day), heart disease (ischemic or congestive), hepatic disease (viral hepatitis, autoimmune hepatitis, wilson disease, hemochromatosis, liver mass lesion), renal disease (serum creatinine concentration of > 1.5 mg/dl), any severe systemic co-morbidities, neoplasm, using any hepatotoxic medication during the past 3 months, previous history of peptic ulcer, previous history of H.pylori eradication, and pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline liver function tests at Twelve weeks | Twelve weeks

SECONDARY OUTCOMES:
Change of insulin resistance and lipid profile during the study period | Twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raika Jamali, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Gastroenterology clinic, Sina Hospital (Tehran) / Beheshti Hospital (Kashan), Tehran / Kashan, Iran